CLINICAL TRIAL: NCT07133802
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Protective Efficacy and Safety of a Nasal Spray Live Attenuated Influenza Vaccine in Adults Aged 18-59 Years
Brief Title: Clinical Trial to Evaluate the Protective Efficacy and Safety of a Nasal Spray Live Attenuated Influenza Vaccine (LAIV) in Adults Aged 18-59 Years Post-Vaccination
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: Hubei Provincial Center for Disease Control and Prevention (Other); Center for Disease Control and Prevention, Fujian (Other); Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B1506-20250113
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Prevention of Influenza

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal Spray Live Attenuated Influenza Vaccine (Experimental)
  Interventions: Biological: Test Group
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo Group

INTERVENTIONS:
Biological: Placebo Group — Each human dose: 0.2 mL
  Arms: Placebo
Biological: Test Group — Each human dose is 0.2 mL
  Arms: Nasal Spray Live Attenuated Influenza Vaccine

SUMMARY:
A Clinical Trial to Evaluate the Protective Efficacy and Safety of a Nasal Spray Live Attenuated Influenza Vaccine (LAIV) in Adults Aged 18-59 Years Post-Vaccination

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged 18-59 years
2. Capable of providing informed consent in person
3. Willing and able to comply with all clinical trial requirements

Exclusion Criteria:

1. Axillary temperature >37.0°C on enrollment day *
2. Received any influenza vaccine within the past 6 months or plans to receive other influenza vaccines during the trial
3. History of laboratory-confirmed influenza (by clinical, serological, or microbiological methods) within the past 6 months
4. Female participants of childbearing potential with positive urine pregnancy test, currently breastfeeding, or planning pregnancy within 6 months
5. Acute phase of any infectious disease/chronic illness within 3 days, or recent use (≤3 days) of antipyretics/analgesics/antihistamines *
6. History of severe allergies requiring medical intervention (e.g., anaphylaxis, angioedema, Arthus reaction) or hypersensitivity to vaccine components (egg proteins, gentamicin sulfate, etc.)
7. Known malignancies, autoimmune diseases (e.g., SLE, rheumatoid arthritis), or immunodeficiency (HIV, organ transplantation, etc.)
8. Asplenia, functional asplenia, or any splenectomy history
9. Use of immunosuppressants/immunomodulators (e.g., systemic corticosteroids >14 days) within 6 months or planned use during study
10. Congenital anomalies affecting organ function, uncontrolled hypertension (≥140/90 mmHg despite treatment), or severe hepatic/renal diseases (e.g., diabetes-complicated)
11. Active asthma or clinical remission for <12 months
12. History or family history of neurological/psychiatric disorders (e.g., epilepsy, Guillain-Barré syndrome)
13. Salicylate use (e.g., aspirin) within 30 days or planned use within 6 weeks post-vaccination
14. Nasal abnormalities potentially affecting vaccine administration (e.g., active allergic rhinitis with medication, ongoing nasal sprays)
15. Blood products/immunoglobulin administration within 3 months or planned use during trial
16. Live-attenuated vaccines within 14 days or subunit/inactivated vaccines within 7 days prior to enrollment *
17. Participation in other clinical trials within 1 month or concurrent involvement in interventional studies
18. Any condition deemed by investigators to compromise trial integrity

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6680 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Protective Efficacy | at 14 days post-vaccination
  To evaluate the protective efficacy of a nasal spray live attenuated influenza vaccine (LAIV) against laboratory-confirmed influenza in participants aged 18-59 years at 14 days post-vaccination

SECONDARY OUTCOMES:
Protective Efficacy | at 14 days post-vaccination
  To evaluate the protective efficacy of a nasal spray live attenuated influenza vaccine (LAIV) against laboratory-confirmed vaccine-matched influenza in participants aged 18-59 years at 14 days post-vaccination
Protective Efficacy | Throughout the entire study period
  To evaluate the protective efficacy of a nasal spray live attenuated influenza vaccine (LAIV) against laboratory-confirmed influenza in participants aged 18-59 years post-vaccination
Protective Efficacy | Throughout the entire study period
  To evaluate the protective efficacy of a nasal spray live attenuated influenza vaccine (LAIV) against laboratory-confirmed, vaccine-matched influenza in participants aged 18-59 years post-vaccination
Safety | 14 days post-vaccination
  Incidence of solicited adverse events (local and systemic) within 14 days post-vaccination
Safety | 30 days post-vaccination
  Incidence of unsolicited adverse events within 30 days post-vaccination
Safety | During the study period
  Incidence of serious adverse events (SAEs) in all participants from vaccination to end of study
Safety | Day 15 post-vaccination
  Viral shedding assessment at Day 3, Day 7, and Day 15 post-vaccination

IPD SHARING:
Plan to Share IPD: No